CLINICAL TRIAL: NCT01113853
Title: Daily Monitoring of Exhaled Nitric Oxide in Asthmatic Patients Stopping Anti-inflammatory Treatment
Brief Title: Daily Monitoring of Exhaled Nitric Oxide in Asthmatic Patients
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: attilio L Boner, Università di Verona
Other Study IDs: AOV 1360
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2007-01

CONDITIONS: Asthma
Keywords: asthma; exhaled nitric oxide; lung function
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous studies have demonstrated that exhaled nitric oxide can be useful to monitor the efficacy of anti-inflammatory treatment as well as to predict a risk of asthma relapse in asthmatic patients.

The aim of the present study is to evaluate the time course of exhaled nitric oxide in mild asthmatic patients, stopping regular treatment with inhaled corticosteroids, if it is possible, in relationship with symptoms and lung function.

DETAILED DESCRIPTION:
All patients were evaluated with pulmonary lung function, exhaled nitric oxide and peak expiratory flow (PEF) and fill in a personal diary for the first two weeks when patients are in treatment; the same evaluation will be made for other four weeks without treatment.

ELIGIBILITY:
Inclusion Criteria:

* mild asthmatic treated with low dose inhaled steroids for whom it has to be considered stop of steroid treatment according to GINA guidelines

Exclusion Criteria:

* age < 5 years
* chronic respiratory diseases

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with asthma visited in the outpatients clinic at University of Verona were invited to participate to the study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-01; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio L Piacentini, MD, Principal Investigator — Universita di Verona
Locations (1):
- Pediatric Department University of Verona, Verona, Verona, Italy